CLINICAL TRIAL: NCT03296475
Title: A Study of the Intra-operative Biomechanics in Complex Abdominal Wall Reconstruction: Do Changes in Abdominal Biomechanics Correlate With Significant Changes in Lung Compliance and Respiratory Function?
Brief Title: Intraoperative Biomechanics in Complex Abdominal Wall Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17/0344
Record Dates: First submitted 2017-09-05; First posted 2017-09-28 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Ventral Hernia; Abdominal Wall Defect
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Intervention Model Description: A single arm prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Midline Ventral Hernia (Experimental): Main inclusion criteria:
  * Patients with midline hernia defects.
  * Patients with either a maximal ventral hernia axial width of greater than 5cm or a loss of domain of greater then 20%.
  * Patients aged ≥ 18 years old.
  * Midline hernias closed in the midline with primary fascial closure with or without mesh augmentation.
  * Midline ventral hernias of VHWG grade 2 or 3.
  Interventions: Procedure: Abdominal Wall Closure Force (N).

INTERVENTIONS:
Procedure: Abdominal Wall Closure Force (N). — This measurement will be recorded for both the right and left anterior rectus sheath. We will measure this force at three anatomical points 1) at the level of the umbilicus and 2) at the halfway point between the pubic symphysis and the xiphisternum and 3) at the point of maximal hernia defect width.

SUMMARY:
Background: A detailed study of the biomechanical changes before and after abdominal wall reconstruction (AWR) has not been performed. Changes in abdominal wall tension and intra-abdominal pressure have physiological consequences on respiratory and cardiology function. AWR surgeons currently do not know if they are applying too much tension when re-aligning the abdominal wall muscles during AWR. Too much tension is likely to cause respiratory and cardiac post-operative complications. The investigators propose to study the perioperative changes in abdominal biomechanics and cardiorespiratory physiology after AWR. In addition, investigators will also analyze the pre-operative patient CT scan to see if there any CT predictors of post-operative cardiorespiratory complications and hernia recurrence. The researchers hypothesize that there is a threshold value or force at which ventral hernias are repaired 'too tight' subjecting the patient to the increased risk of recurrence and cardiorespiratory complications.

Method: An in depth biomechanical and physiological study of 18-22 participants with midline ventral hernias will be carried out. Ventral hernias at least 5cm in width and only those in which primary fascial closure have been achieved will be included. Any operative technique used to achieve primary fascial closure will be included. Biomechanical and physiological measurements will be taken at five separate stages during the course of the patients' abdominal wall reconstruction. The final lung function tests, taken six weeks post op, will be compared to the patients' pre-operative tests. Meticulous attention will be paid to the study protocol making sure that in each patient the measurements are all taken at the same time and under the same conditions.

Discussion: This full biomechanical and physiological work up will enable AWR surgeons to assess when an AWR patient is subjected to too much biomechanical and physiological stress. The abdominal wall tension and strain will be measured to see if this predicts post complications and hernia recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with midline hernia defects. Only patients with one or more midline defect will be included. For our study, we will define a midline hernia as herniation through the linea alba and with the rectus muscles falling either side of the hernia. The pre-operative CT scan will be used to study the hernia morphology and to see whether the patient fulfills these criteria.
* Patients undergoing primary or incisional ventral hernia repair, without formation of or closure of a stoma.
* Patients with either a maximal ventral hernia axial width of greater than 5cm or a loss of domain of greater then 20%, as measured on their pre-operative CT or MRI scan. The loss of domain will be measured using the patients' preoperative CT or MRI scan following the method of Tanaka et al.
* Patients aged ≥ 18 years old.
* Midline hernias closed in the midline with primary fascial closure with or without mesh augmentation. Any reconstruction technique can be used (e.g. anterior or posterior component separation) as long as primary fascial closure is achieved. The mesh may be placed in either the retro-rectus position (with or without a transverse abdominis release) or the onlay position.
* Participants who have a synthetic or bio-synthetic mesh implanted.
* Midline ventral hernias of VHWG grade 2 or 3. Clean and or Clean-contaminated wound classification.
* The participant is legally competent, has been informed of the nature, the scope and the relevance of the study, voluntarily agrees to take part and has duly signed the consent form.

Exclusion Criteria:

* Emergency/Redo surgery.
* Defects not in the midline. Patients with one or more defect not through the linea alba on the pre-operative CT scan.
* AWR for abdominal wall sarcoma, invasive intra-abdominal carcinoma or other malignant disease.
* Contaminated VHWG grade 4 hernias. Or Contaminated or Dirty wound according to the CDC wound classification system.
* Concomitant procedures such as bowel resection.
* The hernia requires a bridged repair.
* Individuals with co-morbid respiratory disease requiring oral corticosteroids or home oxygen therapy.
* Individuals who require the mesh to be placed in the intra-abdominal position.
* A patient with active peritonitis or an active mesh or subcutaneous infection.
* Individuals with a diagnosis of Crohn's disease.
* Individuals of American Society of Anesthesiology grade 4 or 5.
* Complete removal of an existing synthetic mesh (or biosynthetic mesh if not absorb) from a prior hernia repair in the same location is not possible.
* Participants with human immunodeficiency virus (HIV), known liver cirrhosis or alcohol abuse with a known relapse within 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-09 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Dynamic Lung Compliance (measured in ml/cmH2O) | Day 1. Both measurements will be taken on the participants first day of the study. (Study enrollment will take place on the day of the participants operation.
  The primary outcome is the difference in Lung Compliance between stages 3 and 4 of the peri-operative protocol. i.e. we will measure the change in dynamic lung compliance before (after adhesiolysis) and after abdominal wall closure. We will measure this with a standard operative ventilator. Every patient will have a definitive airway (ET tube) fitted.

SECONDARY OUTCOMES:
Perioperative changes in Total Lung Capacity (Litres) | TLC will be measured on Day 1 and at 6 weeks, 12 months and 3 years after the patients operation.
  Total Lung Capacity (TLC) (Litres). TLC will be measured using spirometry before and after the patients AWR operation.
Perioperative changes in Force Expiratory Volume (Litres) | FEV1 will be measured on Day 1 and at 6 weeks, 12 months and 3 years after the patients operation.
  Force Expiratory Volume over 1 second, FEV1 (Litres). FEV1 will be measured using spirometry before and after the patients AWR operation.
Perioperative changes in Tidal Volume (Litres) | VT will be measured on Day 1 and at 6 weeks, 12 months and 3 years after the patients operation.
  Tidal Volume, VT (Litres). VT will be measured using spirometry before and after the patients AWR operation.
Perioperative changes in Residual Volume (Litres) | RV will be measured on Day 1 and at 6 weeks, 12 months and 3 years after the patients operation.
  Residual Volume, RV (Litres). RV will be measured using spirometry before and after the patients AWR operation.
Perioperative changes in Peak Expiratory Flow (Litres/min) | PEF will be measured on Day 1 and at 6 weeks, 12 months and 3 years after the patients operation.
  Peak Expiratory Flow, PEF (Litres/min). PEF will be measured using spirometry before and after the patients AWR operation.
Perioperative changes in Dynamic Lung Compliance (ml/cmH2O) | LC will be measured on Day 1 and at 6 weeks, 12 months and 3 years after the patients operation.
  Dynamic Lung Compliance, LC (ml/cmH2O). LC will be measured using spirometry before and after the patients AWR operation.
Abdominal wall closure force before abdominal wall closure (Newtons) | Day 1. These abdominal wall closure measurements will be taken during the participants operation on the first day of the study. i.e. after enrollment, which will take place on the day of their operation.
  Measured in Newtons (N) with a Mecmesin Newton meter. After adhesiolysis (stage 3) and before abdominal wall closure.
Abdominal wall strain index (no units) (this is a strain index, change in transverse length (cm) / original transverse length of abdominal wall (cm)) | Day 1. Defect width readings taken during the abdominal wall reconstruction operation
  Calculated using the pre-operative CT or MRI and by recording the hernia defect width intra-operatively.
Ventral hernia recurrence | At 1 year after the patients operation.
  Rate of ventral hernia recurrence at 1 year, defined by clinical examination and supplemented by cross-sectional imaging where there is diagnostic uncertainty. Recurrence will be defined using the European classification for ventral hernia recurrence.
Perioperative change in Intra-abdominal pressure (IAP) (mmHg) | Day 1. Readings taken during the abdominal wall reconstruction operation
  Intra-abdominal pressure IAP (mmHg) will be measured using a transducer probe inserted into the bevel of a urinary catheter. The bladder will be inflated with 50ml of normal saline solution, the catheter will be clamped off distal to the position of the transducer/bevel. The bag of normal saline will be lowered to the level of the bladder when the IAP readings are taken. IAP reading will be taken at stages 2, 3 and 4 of our protocol (ie after induction of anaesthetic, after adhesiolysis, and after abdominal wall closure).
Perioperative change in cardiac output (CO) (L/min) | Day 1. Readings taken during the abdominal wall reconstruction operation
  Each participant will be fitted with an oesophageal doppler probe during their operation. This will measure the cardiac output. CO readings will be taken at stages 2, 3 and 4 of our protocol (ie after induction of anaesthetic, after adhesiolysis, and after abdominal wall closure).
Perioperative change in stroke volume (SV) (L) | Day 1. Readings taken during the abdominal wall reconstruction operation
  Each participant will be fitted with an oesophageal doppler probe during their operation. This will measure the cardiac stroke volume. SV readings will be taken at stages 2, 3 and 4 of our protocol (ie after induction of anaesthetic, after adhesiolysis, and after abdominal wall closure).
Perioperative change in positive-end expiratory pressure (PEEP) (cm/H2O) | Day 1. Readings taken during the abdominal wall reconstruction operation
  Positive-end expiratory pressure (PEEP) (cm/H2O) will be measured using the operative ventilator during the patient's operation. PEEP readings will be taken at stages 2, 3 and 4 of our protocol (ie after induction of anaesthetic, after adhesiolysis, and after abdominal wall closure).
Perioperative change in fraction of inspired oxygen (fraction or as a per cent) | Day 1. Readings taken during the abdominal wall reconstruction operation
  Fraction of inspired oxygen (FiO2) will be measured using the operative ventilator during the patient's operation. FiO2 readings will be taken at stages 2, 3 and 4 of our protocol (ie after induction of anaesthetic, after adhesiolysis, and after abdominal wall closure).
Perioperative physiological changes in partial pressure of oxygen (pO2) (kPA) | Day 1. Readings taken during the abdominal wall reconstruction operation
  Blood partial pressure of oxygen (pO2) (kPA) will be measured from arterial gas samples that will be taken from the patients arterial line during the operation.
  pO2 readings will be taken at stages 2, 3 and 4 of our protocol (ie after induction of anaesthetic, after adhesiolysis, and after abdominal wall closure).
Rates of (a) intra-operative, (b) early post-operative (within 30 days of operation) and (c) late post-operative complications. | Up to 3 years after the patients operation.
  Early and late complications will be grouped into local wound complications (e.g. wound infection, seroma etc) and systemic complications (e.g. pneumonia, myocardial infarction etc). We will follow the Clavien-Dindo classification scheme.
Ventral hernia recurrence | At 3 year after the patients operation.
  Rate of ventral hernia recurrence at 3 years, defined by clinical examination and supplemented by cross-sectional imaging where there is diagnostic uncertainty. Recurrence will be defined using the European classification for ventral hernia recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Emerton, BA, Study Director — Joint Research Office, University College London
Locations (1):
- Univeristy College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Designated members of the research team will be responsible for data entry at different steps of the patient pathway. All researchers will be responsible for the accuracy of the documentation and must ensure that all entries can be verified by the source data. An explanation will be given for all missing data. All the study documents and proformas containing the participant data will be kept on site in the General Surgery department at our hospital. At no point, will these documents be removed from the department. Study data will be pseudo-anonymised for data analysis. The file containing the pseudo-anonymised data will be password protected. Only the pseudo-anonymised data will leave the hospital department, it will be transferred using the secure UCLH.nhs.uk and NHS.net email systems. Only the primary researcher, SGP, will have access to the pseudo-anonymised data outside our hospital department, where the password protected data file will be keep on his secure personal laptop.